CLINICAL TRIAL: NCT01518452
Title: Computerized Working Memory Training Evaluated With Clinical Assessments and Quantitative EEG in Very-low-birth-weight (VLBW) Children at Preschool Age
Brief Title: Computerized Working Memory Training in Very-low-birth-weight Children at Preschool Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/532
Record Dates: First submitted 2012-01-10; First posted 2012-01-26 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Infant, Very Low Birth Weight
Keywords: working memory training, computerized; clinical assessment; quantitative EEG; child, preschool

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- working memory training (Experimental): Cogmed JM working memory training
  Interventions: Behavioral: Cogmed JM working memory training
- delayed working memory training (Experimental): Cogmed JM working memory training after 8 weeks waiting
  Interventions: Behavioral: Cogmed JM working memory training after waiting

INTERVENTIONS:
Behavioral: Cogmed JM working memory training — daily training for 5 weeks on a computerized program for training working memory; a total of 25 training sessions. Program: Cogmed JM - preschool version of program: 15-20 minutes training per day
  Arms: working memory training
Behavioral: Cogmed JM working memory training after waiting — Waiting after baseline testing for 8 weeks. Daily training on a computerized program for training working memory for 5 weeks. 25 training sessions in total. Program: Cogmed JM - preschool version of program: 15-20 minutes training per day
  Arms: delayed working memory training

SUMMARY:
The main aim of this prospective interventional study is to compare quantitative EEG findings and cognitive and neuropsychological test results before and after training with the Cogmed JM program in a group of very-low-birth-weight children in preschool age, i.e. ages 5-6 years. The investigators hypothesize that the children in the study may respond positively to the computerized training and improve working memory, but probably to different degrees depending on the underlying neurological condition. The investigators also hypothesize that training may benefit additional executive functions.

DETAILED DESCRIPTION:
Children born preterm are at increased risk of neurological disabilities due to perinatal brain damage. During the last ten years an increasing number of especially extremely low birth weight (ELBW: BW ≤ 1000g) children has survived, and one might wonder whether this has lead to increased amount of brain pathology and impairments among survivors. Major impairments including cerebral palsy, mental retardation and impaired vision and hearing are most common in children born extremely preterm (gestational age below 28 weeks). In addition to this, a large part of survivors after preterm birth will experience motor problems, cognitive dysfunctions, psychiatric and behavioural problems of varying severity.

In our previous research we have found significant deficits in working memory in very preterm born children, and this seems to have a strong influence on cognitive functioning. During the last years, several studies have shown that working memory skills can be trained, and training working memory to improve cognition and executive functions is regarded as one of the major steps forward in neuroscience in recent years.

The working memory training program version for preschoolers, Cogmed JM, has recently been launched. Healthy preschoolers trained on working memory improved significantly on trained tasks but also on non-trained tests of spatial and verbal working memory, as well as transfer effects on attention. The preschool version of the program has not yet been administered to preterm born or other neurologic high risk children in this age group.

The main aim of this prospective interventional study is to compare quantitative EEG findings and cognitive and neuropsychological test results before and after training with the Cogmed JM program in a group of very-low-birth-weight children in preschool age, i.e. ages 5-6 years. We hypothesise that the children in the study may respond positively to the computerized training and improve working memory, but probably to different degrees depending on the underlying neurological condition. We also hypothesise that training may benefit additional executive functions.

The children in the study will be divided into two subgroups (15/15 children). Subgroup A will start training, while subgroup B waits during this first training period. Subgroup B will therefore act as a control group. After 8 weeks subgroup B will then start training. This is in agreement with the so-called Stepped Wedge design (Brown and Lilford 2006).

ELIGIBILITY:
Inclusion Criteria:

* VLBW (birth weight ≤ 1500 grams)
* preschool child
* born at St. Olav's University Hospital in Trondheim in 2005 and 2006

Exclusion Criteria:

* birth weight >1500 grams
* diagnosed genetic syndromes
* severe cerebral palsy with totally impaired bilateral hand function (GMFCS - gross motor function classification scale level V)
* blindness

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
working memory capacity | 6 months
  Automated Working Memory Assessment (AWMA)(visual working memory); digit span (from WISC-IV); Repetition of scentences (from NEPSY battery); Remembering and oral story (from NEPSY battery); Remembering faces (from NEPSY battery)

SECONDARY OUTCOMES:
behavioral function | 6 months
  Vineland adaptive behaviour scales (survey form)
executive function | 6 months
  The ADHD Rating Scale-IV (parents report)
anxiety as judged by parents | 6 months
  The Screen for Child Anxiety Related Emotional Disorders (SCARED- parent report); Preschool Anxiety Scale (parent report)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Skranes, PhD prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Grunewaldt KH, Lohaugen GC, Austeng D, Brubakk AM, Skranes J. Working memory training improves cognitive function in VLBW preschoolers. Pediatrics. 2013 Mar;131(3):e747-54. doi: 10.1542/peds.2012-1965. Epub 2013 Feb 11. PMID 23400616
- [Result] Grunewaldt KH, Skranes J, Brubakk AM, Lahaugen GC. Computerized working memory training has positive long-term effect in very low birthweight preschool children. Dev Med Child Neurol. 2016 Feb;58(2):195-201. doi: 10.1111/dmcn.12841. Epub 2015 Jul 3. PMID 26140426